CLINICAL TRIAL: NCT00382122
Title: Prevalence of Ocular Surface Disease in Glaucoma Patients
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: CMS-06-06
Record Dates: First submitted 2006-09-27; First posted 2006-09-28 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2007-09

CONDITIONS: Glaucoma
Keywords: Glaucoma; Ocular hypertension; Dry eye; Ocular surface disease
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Demographic information and a brief medical and concomitant medicine history will be obtained from the glaucoma patient's records. Qualified patients will be asked to complete a questionnaire about their symptoms. Patients will then be scheduled to undergo three standard clinical tests of the ocular surface.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glaucoma;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Inability to understand trial procedures;
* Inability to understand Informed Consent;
* Current use or use within the last 3 months of Restasis, steroids, or topical ocular non-steroidal anti-inflammatory drugs;
* Punctal plugs;
* Previous glaucoma, corneal, or conjunctival surgery;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older with open-angle glaucoma or ocular hypertension were consecutively recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2006-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Medeiros, MD, PhD, Study Director — University of California, San Diego
Locations (1):
- La Jolla, La Jolla, California, United States

REFERENCES:
- [Result] Leung EW, Medeiros FA, Weinreb RN. Prevalence of ocular surface disease in glaucoma patients. J Glaucoma. 2008 Aug;17(5):350-5. doi: 10.1097/IJG.0b013e31815c5f4f. PMID 18703943